CLINICAL TRIAL: NCT00292292
Title: Clinical Study Protocol for the Investigation of the Kineflex Spinal System - a Pivotal Study in Continued Access Stage
Brief Title: Kineflex Artificial Disc System to Treat Degenerative Disc Disease (DDD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Economic and business reasons
Sponsor: SpinalMotion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kineflex
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-08

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kineflex Lumbar Artificial Disc (Experimental): Treatment arm
  Interventions: Device: Lumbar Artificial Disc
- Charite (Active Comparator)
  Interventions: Device: Charite Artificial Disc

INTERVENTIONS:
Device: Lumbar Artificial Disc — Insertion of the Kineflex Lumbar ArtificialDisc
  Other Names: Kineflex Disc
  Arms: Kineflex Lumbar Artificial Disc
Device: Charite Artificial Disc — Insertion of the Charite
  Other Names: SB Charite
  Arms: Charite

SUMMARY:
The Kineflex Spinal System is no worse than the Charite Spinal System in patients with single level degenerative disc disease at L4/5 or L5/S1.

DETAILED DESCRIPTION:
The Kineflex disc is a 3-piece modular design consisting of 2 cobalt chrome molybdenum (CCM) end-plates and a fully articulating CCM core. The system is available in 3 foot print sizes.

ELIGIBILITY:
Inclusion Criteria Summary:

* Be between 18 and 60 years of age
* Have evidence of degenerative disc disease (DDD)
* History of back and/or radicular pain which is severe, ongoing and recurrent
* Minimum 6 month period of prior conservative care
* Moderate Oswestry Disability Index score
* Moderate pain score
* Be likely to return for all follow-up visits
* Be willing and able to provide Informed Consent for study participation.

Exclusion Criteria Summary:

* Any back or leg pain of unknown origin
* Foot drop
* Previous trauma to the study treatment level with compression or bursting
* Previous retroperitoneal surgery
* Other spinal surgery at affected level except IDET, laminotomy
* Previous thoracic or lumbar fusion
* Documented abnormal abdominal vessel or muscular/fascial pathology or morphology
* Degenerative spondylolisthesis
* Ischemic (spondylolytic) spondylolisthesis
* Spondylitis
* Documented significant spinal, foraminal or lateral stenosis
* Severely reduced disc space height
* Documented presence of free nuclear fragment
* Extensive facet arthritis or degeneration of the facets at any level noted on MRI, CT or X-ray
* Scoliosis of the lumbar spine
* Metabolic bone disease
* Active systemic infection
* Hepatitis
* Active malignancy or history of metastatic malignancy
* Any terminal or autoimmune disease
* Any other disease, condition or surgery which might impair healing
* Recent history of chemical or alcohol dependence
* Current or extended use of any drug known to interfere with bone or soft tissue healing
* Known metal allergy
* Morbid obesity
* Transitional vertebrae at level to be treated that has not clearly fused
* Currently a prisoner
* Currently involved in spinal litigation
* Currently experiencing an episode of major mental illness
* Pregnancy at time of enrollment, since this would contraindicate abdominal surgery
* Participation in another drug, diologic or medical trial within 30 days of study surgery
* Lives more than 300 miles from a study center or participation in any other investigational drug, biologic or medical device study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 514 (Actual)
Dates: Start 2005-01; Primary Completion 2009-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Improvement in Oswestry Low Back Pain Disability Score at 24 months compared with baseline; no revision removal, supplemental fixation or device related reoperations and no major adverse event as defined by the study protocol | 24 months

SECONDARY OUTCOMES:
Maintenance or improvement in neurologic status | 24 months
Pain improvement | 24 months
Significant disc height increase | 24 months
No displacement or migration of the device | 24 months
Time to return to work | 24 months
Time to recovery | 24 months
Preservation of at least 4 degrees of motion in flexion/extension | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Fred Geisler, MD, Principal Investigator — Medical Monitor
Locations (21):
- United States (21):
  - Tower Orthopedics and Sports Medicine, Beverly Hills, California
  - CORE Orthopaedic Medical Center, Encinitas, California
  - Kaiser Oakland Regional Spine Surgery, Oakland, California
  - Loma Linda University, San Bernardino, California
  - University of California San Diego, San Diego, California
  - UCSF Dept. of Orthopaedic Surgery, San Francisco, California
  - Rocky Mountain Associates in Orthopedic Medicine, P.C., Loveland, Colorado
  - Illinois Neuro-Spine Center, Aurora, Illinois
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Maryland Brain and Spine Center, Annapolis, Maryland
  - Orthopaedic Associates, P.A, Towson, Maryland
  - Sierra Regional Spine Institute, Reno, Nevada
  - Hamilton Orthopaedic Surgery and Sports Medicine, Hamilton, New York
  - Buffalo Spine Surgery, Lockport, New York
  - Manhattan Orthopaedics, P.C., New York, New York
  - Carolina Neurosurgery and Spine Associates, Charlotte, North Carolina
  - Triangle Orthopaedic Associates, P.A., Durham, North Carolina
  - Univ. of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Texas Back Institute Clinical Research Organization, Plano, Texas
  - Gordon Spine Associates, Tyler, Texas
  - Orthopedics International Spine, Kirkland, Washington

REFERENCES:
- See also: sponsors web site contains animated information regarding disc — http://www.spinalmotion.com